CLINICAL TRIAL: NCT00648557
Title: Single-Dose Fasting In Vivo Bioequivalence Study of Levothyroxine Sodium Tablets (200 mg; Mylan) to Synthroid Tablets (200 mg; Abbott) in Healthy Volunteers
Brief Title: Fasting Study of Levothyroxine Sodium Tablets 200 mg to Synthroid Tablets 200 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LEVO-02144
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Thyroxine

ARMS (2):
- 1 (Experimental): Levothyroxine Sodium Tablets 200 mg
  Interventions: Drug: Levothyroxine Sodium Tablets 200 mg
- 2 (Active Comparator): Synthroid Tablets 200 mg
  Interventions: Drug: Synthroid Tablets 200 mg

INTERVENTIONS:
Drug: Levothyroxine Sodium Tablets 200 mg — 3x200mcg, single dose fasting
  Arms: 1
Drug: Synthroid Tablets 200 mg — 3x200mcg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's levothyroxine sodium 200 μg tablets to Abbott's Synthroid® 200 μg tablets following a single 600 μg (3 x 200 μg) dose administration in healthy volunteers under fasting conditions. Twenty-nine healthy, non-smoking, subjects between the ages of 18 and 47 completed this open-label, randomized, two-period, two-treatment, single-dose crossover study conducted by Dr. James D. Carlson at PRACS Institute, Ltd., Fargo, ND. Statistical analysis of the data revealed that 90% confidence intervals were within the acceptable bioequivalent range of 80% and 125% for the natural log transformed parameters LNAUC0-48hr and LNCPEAK for baseline corrected total L-thyroxine. This study demonstrated that Mylan's 200 μg levothyroxine sodium tablets are bioequivalent to Abbott's Synthroid® 200 μg tablets following a single, oral 600 μg (3 x 200 μg) dose under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-50 years.
2. Sex: Men and/or non-pregnant, non-lactating women.

   1. Women of childbearing potential must have negative serum β human chorionic gonadotropin (HCG) pregnancy tests performed within 14 days prior to of the study and on the evening prior to each dose administration. An additional serum (β HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or be using an acceptable form of contraception throughout the duration of the study. Oral contraceptives are not to be used within 3 months prior to dosing and throughout the course of the study due to the fact that they increase serum TBG concentrations, and therefore, elevate T4. Acceptable forms of contraception include the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. postmenopausal accompanied with a documented postmenopausal course of at least one year or surgical sterility (tubal ligation, oophorectomy or hysterectomy).
3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women, and within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1983 (See Part II Administrative Aspects of Bioequivalence Protocols).
4. All subjects should be judged normal (euthyroid) and healthy during a prestudy medical evaluation (physical examination, laboratory evaluation, blood chemistry, serum T4 (free and total), serum T3 (total only), serum thyroid-stimulating hormone (TSH), serum thyroxine-binding globulin (TBG), hepatitis B and hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepine, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the initial study drug administration.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins within the 48 hours prior to the initial dose of the study medication.
   4. Any change in dietary or exercise habits throughout the duration of the study.
3. Medications:

   1. Use of any medication within the last 30 days prior to the initial dose of study medication, during the study or during the washout period. These may include but is not limited to: infant soybean formula, steroids, salicylates, androgenic or estrogenic hormones including oral contraceptives; preparations containing iodine, such as vitamins; oral anti-diabetic agents; all resins for lowering of cholesterol, such as cholestyramine; sucralfate, propranolol, amiodarone, phenytoin, carbamazepine, furosemide; aluminum-containing antacids, including aluminum hydroxide; rifampin, calcium channel blockers and ferrous sulfate.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant chronic disease and/or hepatitis.
   2. History of drug and/or alcohol abuse.
   3. Acute illness at the time of either the prestudy medical evaluation or dosing.
   4. History of any thyroid disease.
   5. Subjects with any underlying medical condition known to interfere with the absorption or metabolism of thyroid hormones.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide for Clinically Relevant Abnormalities (See Part II Administrative Aspects of Bioavailability Protocols).
   2. Abnormal and clinically relevant ECG tracing.
   3. Abnormal thyroid function tests.
6. Donation or loss of a significant volume of blood or plasma (> 450 ml) within 28 days prior to the initial dose of study medication.
7. Subjects who received any surgical treatment within 6 months prior to the initial dose of study medication.
8. Subjects with known allergies or hypersensitivity to thyroid preparations.
9. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2003-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html